CLINICAL TRIAL: NCT04615442
Title: ECV - Epihunter Clinical Validation
Acronym: ECV
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Epihunter NV (Industry)
Collaborators: Filadelfia Epilepsy Hospital (Other); KU Leuven (Other); Boston Children's Hospital (Other); Institute of Neurology and Neuropsychology, Tbilisi, Georgia (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: EPI2019B
Record Dates: First submitted 2020-09-14; First posted 2020-11-04 (Actual); Last update posted 2022-04-04 (Actual); Status verified 2022-04

CONDITIONS: Absence Seizures; Absence Epilepsy
MeSH Terms: conditions — Seizures; Epilepsy, Absence

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- All subjects (Experimental): Subjects that undergo a clinical video EEG are asked to additionally wear a wearable EEG headband for up to 2 periods of 4h during the video EEG.
  Interventions: Device: Epihunter

INTERVENTIONS:
Device: Epihunter — Subjects wear epihunter during routine video EEG

SUMMARY:
The goal of this prospective study is to validate a wearable EEG seizure detection solution compared to video EEG. Subjects that undergo a clinical video EEG are asked to additionally wear a wearable EEG headband for up to 2 periods of 4h during the video EEG.

ELIGIBILITY:
Inclusion Criteria:

* Subjects should have an indication of having absence seizures
* Subjects should be admitted for video EEG monitoring as part of their clinical practice
* Age > 4 years

Exclusion Criteria:

* Head circumference should be compatible for wearable EEG device (40-70cm)
* The subject should be able to understand instructions and refrain from removing the device from its head

Min Age: 4 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 102 (Actual)
Dates: Start 2020-05-01 (Actual); Primary Completion 2021-06-28 (Actual); Study Completion 2021-12-31 (Actual)

PRIMARY OUTCOMES:
Sensitivity for electrographic seizures of study device compared to video EEG | 9 months
  The sensitivity for electrographic seizures by the study device compared to manually annotated electrographic seizures on non-video EEG is > 0.90 (median sensitivity per patient)
Number of false alarms by study device per hour | 9 months
  The number of false alarms by the study device < 0.1 per hour (median false detection rate per recording)

SECONDARY OUTCOMES:
Feasibility testing of automated behavioral testing triggered by automated detection | 3 months
  Assess if automated behavioral testing triggered by automated detection can be used to automatically assess awareness during an absence seizure. Successful if subjects DO NOT react to the testing during an unaware seizure, and DO react during an aware seizure.

CONTACTS AND LOCATIONS:
Overall Officials: Dirk Loeckx, PhD, Principal Investigator — Epihunter NV
Locations (4):
- Boston Children's Hospital, Boston, Massachusetts, United States
- UZ Leuven, Leuven, Belgium
- Danish Epilepsy Center, Dianalund, Denmark
- Institute of Neurology and Neuropsychology, Tbilisi, Georgia